CLINICAL TRIAL: NCT05811936
Title: A Randomized Controlled Trial to Evaluate the Survivorship Needs Assessment Planning (SNAP) Tool for Head and Neck Cancer Survivor-Caregiver Dyads
Brief Title: The SNAP Tool for Head and Neck Cancer Survivor-Caregiver Dyads
Acronym: SNAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Katherine Sterba, Professor • COM PHS Administration CC, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 00114288; R01CA259186-01 (NIH); R01CA259186-02 (NIH)
Record Dates: First submitted 2023-03-15; First posted 2023-04-13 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Cancer; Survivorship; Caregiver Burden; Head and Neck Neoplasms
Keywords: Head and Neck Cancer; Survivorship
MeSH Terms: conditions — Head and Neck Neoplasms; Caregiver Burden | interventions — Equipment and Supplies

STUDY DESIGN:
Intervention Model Description: Patient and Caregiver dyads will be randomized to either the SNAP intervention group or the Usual Care (UC) group after baseline assessment. Dyads will be randomized to study arm (SNAP or UC) using permuted block randomization with block sizes of 2 or 4. Randomization will be stratified by patient gender (male or female) and treatment (radiation only, radiation + surgery OR chemotherapy, radiation + surgery + chemotherapy).
Masking Description: Study personnel (Coordinator, Nurse, Data Collectors) will not be blinded to group as intervention activities differ by group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention): Caregiver- Survivor Dyads in this group will receive routine follow-up care in the HNC clinic. Current standard of care is an Advanced Practice Provider (Physician Assistant or Nurse Practitioner)-delivered survivorship visit after treatment. This visit will take place according to UC in the clinic. UC dyads will also receive printed caregiving and survivorship materials.
- SNAP (Experimental): Caregiver- Survivor Dyads in this group will receive a two-session intervention spanning 3 months, with a caregiver module within 1-2 weeks of the end of RT and a dyadic module at 3 months. Each session will include a needs- assessment, a tailored care plan with a goal setting discussion, and referrals for unmet needs. Each session follows with a supportive mobile app for 6 weeks.
  Interventions: Behavioral: Survivorship Needs Assessment Planning (SNAP) tool

INTERVENTIONS:
Behavioral: Survivorship Needs Assessment Planning (SNAP) tool — SNAP includes 2 educational survivorship modules for caregivers and survivors. There are 3 main elements: needs assessment, a tailored care plan and a mobile support app. SNAP uses pre-specified categories of needs, resources, and messaging "behind the scenes" to automate the identification, rating and management of high priority needs. Generated tailored care plans include referrals, messages and educational materials mapped to prioritized dyad-reported concerns addressing survivorship domains (diagnosis, treatment, follow-up care). Care plans and referrals are reviewed with an Advanced Practice Provider. Barriers to uptake are addressed, goal-oriented action planning is refined with brief mobile app training. Dyads receive a personalized binder with care plan, referrals, and an action plan. Dyads receive e-monitoring for 6 weeks to check in and identify barriers with algorithm-driven messaging to reinforce progress, provide further resources and encouragement.
  Other Names: SNAP
  Arms: SNAP

SUMMARY:
In this randomized behavioral intervention, head and neck cancer (HNC) survivors and their caregivers (N=176 HNC survivor-caregiver dyads) will be randomized to either Survivorship Needs Assessment Planning (SNAP) or Usual Care (UC) groups to examine the effects of SNAP on outcomes. SNAP includes two sessions with a needs assessment and tailored care plan and a supportive mobile app after completion of radiation to promote uptake of recommended medical and supportive care. The study aims to evaluate the effects of SNAP on symptom severity in patients and caregiver burden in caregivers. Secondary outcomes include psychological distress (anxiety and depression), healthcare utilization (receipt of recommended care) and unmet needs and self-efficacy in HNC survivor-caregiver dyads. Participants will complete surveys at baseline, 6 months, and 9 months post randomization with validated PROMs, and receive intervention modules at the end of radiation and month 3. Participants in the SNAP group will also receive mobile app support.

DETAILED DESCRIPTION:
The SNAP Intervention includes two care planning modules, a caregiver visit (module I) during the end of radiation treatment and a dyad-focused (survivor and caregiver) visit (module II) at 3 months. Each SNAP module includes 3 components including: 1) an in-clinic needs assessment, 2) a tailored care plan and 3) text-based e-monitoring at home. In both modules, a care plan is generated with algorithm-triggered messages and referrals to recommended care matched to endorsed concerns. Care plans are reviewed and barriers are addressed. Referrals are finalized with an Advanced Practice Provider (APP). SNAP Participants leave with a personalized binder including the survivorship care plan and referrals. SNAP Participants use an e-monitoring App and receive twice weekly engagement prompts for 6 weeks. Usual Care (UC) participants will receive caregiver education and dyadic survivorship education visit at the end of radiation treatment and 3-months post-randomization, respectively, with printed materials from the National Cancer Institute.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Age >18
2. Stage I-IV non-metastatic HNC (i.e., lip/oral cavity, nasopharynx, salivary gland, oropharynx, hypopharynx, paranasal sinus, larynx and cutaneous cancers)
3. Currently receiving radiation treatment (with/without surgery and/or concurrent chemotherapy) with curative intent
4. Able to nominate caregiver, the primary support person, also interested in participating

Caregiver Inclusion Criteria:

1. Age >18
2. Provide care for a loved one with stage I-IV HNC
3. Agrees to participate after being nominated

Patient Exclusion Criteria:

1. Patients who do not read/understand English
2. Patients who are cognitively impaired and cannot complete interviews as judged by the referring health care provider
3. Patients concurrently diagnosed with and/or receiving treatment for a second "significant" primary cancer, except the following:

   * Excised and cured non-melanoma skin cancer
   * Carcinoma in situ of breast or cervix
   * Superficial bladder cancer
   * Stage 1 differentiated thyroid cancer that is resected or observed
   * pT1a/pT1b prostate cancer comprising <5% of resected tissue with normal prostate specific antigen (PSA) since resection
   * cT1a/cT1b prostate cancer treated with brachytherapy

Caregiver Exclusion Criteria:

1. Inability to read or understand English
2. Cognitively impaired and cannot complete interviews, as judged by the referring health care provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Caregiver Burden at 9 months post randomization | Caregivers will be assessed at baseline, 6 weeks, 6 months, and 9 months post randomization
  Caregivers report the extent to which caregiving impacts time, responsibilities, and strain utilizing the Zarit Burden Inventory. Caregivers rate each item on a 5-point Likert scale (0=Never to 4=Always); higher scores (0-16) indicate greater burden. An increase in change from baseline to 6 week, 6 months or 9 months follow up visit would increased caregiver distress; likewise a decrease in change would indicate reduced caregiver distress. Cronbach's alphas in previous research range from 0.81-0.83.
Change from baseline in Symptom Severity in head and neck cancer survivors at 9 months post randomization | Survivors will be assessed at baseline, and at 6 months and 9 months post randomization
  Symptom burden in survivors will be assessed with the MD Anderson Symptom Inventory-Head and Neck Cancer Module (MDASI-HN) The MDASI -HN includes 13 core items and an additional 9 head and neck cancer module items which calculates a total score of symptom severity. The MDASI assesses the severity of symptoms at their worst in the last 24 hours on a 0-10 Numeric Rating Scale, with 0 being "not present" and 10 being "as bad as you can imagine." Core items and module symptom items are averaged into a mean module severity. A higher score always indicates an increase in severity. A decrease in change from baseline to 9-month assessment indicates improvement of symptoms. Cronbach's alphas in previous research range from 0.88-0.92.

SECONDARY OUTCOMES:
Change from baseline in Depression for Caregivers at 9 months post randomization | Caregivers will be assessed at baseline, 6 months and 9 months
  Depression in Caregivers will be assessed with the PROMIS Depression- SF v1.0 form 8A. Respondents are asked how often in the past 7 days they have experienced specific depression symptoms, using a 5-point ordinal rating scale whereby 1= "Never," 5="Always." A higher score indicates higher depression. Raw score totals are converted to an item response theory-based T-scores. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10 with a range of 38.2 to 81.3. Therefore, a person with a T-score of 40 is one SD below the mean. A decrease in change from baseline to 9 month assessment indicates reduced depression. Cronbach's alphas in previous research = 0.97 for anxiety and depression.
Change from baseline in Anxiety for Caregivers at 9 months post randomization | Caregivers will be assessed at baseline, 6 months and 9 months
  Anxiety in Caregivers will be assessed with the PROMIS Short Form v1.0 - Anxiety 8a. Respondents are asked how often in the past 7 days they have experienced specific anxiety symptoms, using a 5-point ordinal rating scale whereby 1= "Never," 5="Always." A higher score indicates higher anxiety. Raw score totals are converted to an item response theory-based T-scores. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10 with a range of 38.2 to 81.3. Therefore, a person with a T-score of 40 is one SD below the mean. A decrease in change from baseline to 9 month assessment indicates reduced anxiety. Cronbach's alphas in previous research = 0.97 for anxiety and depression.
Change from baseline in Depression for Survivors at 9 months post randomization | Survivors will be assessed at baseline, 6 months and 9 months
  Depression in Survivors will be assessed with the PROMIS Depression- SF v1.0 form 8A . Respondents are asked how often in the past 7 days they have experienced specific depression symptoms, using a 5-point ordinal rating scale whereby 1= "Never," 5="Always." A higher score indicates higher depression. Raw score totals are converted to an item response theory-based T-scores. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10 with a range of 38.2 to 81.3. Therefore, a person with a T-score of 40 is one SD below the mean. A decrease in change from baseline to 9 month assessment indicates reduced depression. Cronbach's alphas in previous research = 0.97 for anxiety and depression.
Change from baseline in Anxiety for Survivors at 9 months post randomization | Survivors will be assessed at baseline, 6 months and 9 months
  Anxiety in Survivors will be assessed with the PROMIS Short Form v1.0 - Anxiety 8a. Respondents are asked how often in the past 7 days they have experienced specific anxiety symptoms, using a 5-point ordinal rating scale whereby 1= "Never," 5="Always." A higher score indicates higher anxiety. Raw score totals are converted to an item response theory-based T-scores. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10 with a range of 38.2 to 81.3. Therefore, a person with a T-score of 40 is one SD below the mean. A decrease in change from baseline to 9 month assessment indicates reduced anxiety. Cronbach's alphas in previous research = 0.97 for anxiety and depression.
Change in Healthcare Utilization (HCU)/ receipt of recommended care at 6 months in head and neck cancer survivor-caregiver dyads. | Dyads (Survivor & Caregiver) will be assessed at baseline, 6 months and 9 months
  Healthcare utilization (HCU) in survivors and caregivers is the receipt of recommended care assessed by self-report and chart review. HCU will be evaluated based on the number of completed referrals dived by the number of recommended medical or supportive care referrals. We will use count-based regression to model the logarithm of the expected number of completed referrals as a function of treatment group with an offset equal to the logarithm of the total number of patient referrals, and baseline covariate adjustment. Based on the fitted model, we will construct point and interval estimates of the rate of HCU for SNAP and UC (Usual Care) dyads. The significance of the intervention on HCU will be based on the statistical significance of the treatment effect parameter. Primary analyses will use chart review data and additional exploratory analyses will use self-reported data.
Change in from baseline Unmet Needs at 6 months in head and neck cancer Caregivers | Caregivers will be assessed at baseline, 6 weeks, 6 months, 9 months
  Unmet needs will be assessed by the Cancer Survivor Partner Unmet Needs (CaSPUN) instrument. Respondents rate 30 items concerning whether they currently needed help with comprehensive care, information, quality of life, existential survivorship and relationship issues (yes or no). Total number of unmet needs will be calculated. Cronbach's alphas in previous research range from 0.93-0.94.
Change in from baseline Unmet Needs at 6 months in head and neck cancer Survivors | Survivors will be assessed at baseline, 6 months, 9 months
  Unmet needs will be assessed by the Cancer Survivor Unmet Needs (CaSUN) instrument. Respondents rate 30 items concerning whether they currently needed help with comprehensive care, information, quality of life, existential survivorship and relationship issues (yes or no). Total number of unmet needs will be calculated. Cronbach's alphas in previous research range from 0.93-0.94.
Change in from baseline Self-efficacy at 6 months in head and neck cancer Caregivers | Caregivers will be assessed at baseline, 6 weeks, 6 months, 9 months
  Caregiver self-efficacy will be assessed with the 21-item Caregiver Inventory measure. Participants will rate the extent to which they feel confident in their abilities as a caregiver to manage medical information, care for their loved one with cancer, manage emotions and care for oneself on a 9 point response scale from not at all confident to totally confident. Higher scores reflect higher self-efficacy (Cronbach's alpha in previous research = 0.91).
Change in from baseline Self-efficacy at 6 months in head and neck cancer Survivors | Survivors will be assessed at baseline, 6 months, 9 months
  Survivor self-efficacy will be assessed with the 12-item Communication and Attitudinal Self-Efficacy Scale (CASE) instrument. Participants will rate the extent to which they feel confident in understanding and participating in their care, maintaining a positive attitude, and seeking and obtaining information on a 4 point response scale from Strongly Disagree (1) to Strongly Agree (4). Higher scores reflect higher self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine R Sterba, PhD, MPH, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No